CLINICAL TRIAL: NCT02234128
Title: A Phase 2, Multicenter, Open-label Study to Measure the Safety of Extending Preservation and Assessment Time of Donor Lungs Using Normothermic Ex Vivo Lung Perfusion and Ventilation (EVLP) as Administered by the SPONSOR Using the Toronto EVLP System™
Brief Title: Extending Preservation and Assessment Time of Donor Lungs Using the Toronto EVLP System™ at a Dedicated EVLP Facility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lung Bioengineering Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PXUS-14-001; 4766 (Other: Sterling IRB)
Record Dates: First submitted 2014-09-04; First posted 2014-09-09 (Estimated); Results first posted 2020-10-09 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Lung Disease
Keywords: Ex Vivo Lung Perfusion; EVLP; Lung Transplant; Lung Transplantation; Toronto EVLP System™; PERFUSIX
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- EVLP Double Lung Group (Experimental): Toronto EVLP System™ administered to double lungs.
  Interventions: Device: Toronto EVLP System™
- EVLP Single Lung Group (Experimental): Toronto EVLP System™ administered to single lungs.
  Interventions: Device: Toronto EVLP System™
- Control Group (No Intervention): Those patients receiving a single or double lung via conventional transplant.

INTERVENTIONS:
Device: Toronto EVLP System™ — Extending preservation and assessment time of donor lungs using the Toronto EVLP System
  Arms: EVLP Double Lung Group; EVLP Single Lung Group

SUMMARY:
This is a safety study to compare the safety of receiving a lung treated with the Toronto EVLP System™ by SPONSOR in SPONSOR's dedicated facility against standard lung transplantation.

DETAILED DESCRIPTION:
Human donor lungs allocated to a participating study transplant center (Study Center) for a specific recipient and meeting study EVLP donor lung inclusion/exclusion criteria will be assessed by SPONSOR for inclusion into the study.

Upon retrieval, donor lung(s) will be packaged and transported on ice to the SPONSOR's EVLP facility in Silver Spring, Maryland, no differently than when lungs are recovered, packaged, and transported to any transplant center for implantation.

The EVLP procedure will be performed by Certified Ex Vivo Lung Specialists using the Toronto EVLP System™ for up to 6 hours, collecting and relaying lung function assessment data hourly or as requested by the Study Center transplant surgeon. Additionally, the Study Center surgeon will have the capability to evaluate lung function data and monitor the procedure remotely through a dedicated video link.

Upon acceptance of an EVLP donor lung by the Study Center, the single lung or lung block is cooled down by the Toronto EVLP System™ to 10 degrees C. Thereafter, perfusion and ventilation are stopped and the lung is prepared for hypothermic storage and transport to the accepting Study Center.

ELIGIBILITY:
Subject Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Male or female patients
* All patients, 18 years of age or older
* Patient already on or added to the active waiting list for a single or bilateral lung transplant
* Patient or patient's representative provides informed consent for participation in the study at the time of study commencement or time of listing for transplant
* Patient or patient's representative reconfirms informed consent for the study on the day of lung transplant

Subject Exclusion Criteria:

A subject who meets any of the following criteria will be excluded from participation:

* Patients listed for same-side lung re-transplantation
* Patients listed for multiple organ transplantation including lung and any other organ
* Patients listed for live donor lobar transplant
* Patients with HIV, active Hepatitis B/C, or Burkholderia Cepacia
* Patients not initially consented into the study prior to the time of lung transplant
* Patients in the ICU at the time of initial lung offer requiring mechanical ventilation, ECMO or other Extracorporeal life support (ECLS).

Donor Lung Inclusion Criteria for EVLP Assessment:

The donor lung must meet at least one of the following criteria to proceed with EVLP:

* At the time of the clinical evaluation, the donor PaO2/FiO2 < 300 mmHg
* Donor received ≥ 10 units of blood transfusions
* Donation after Cardiac Death (DCD) donor
* Expected cold ischemic time > 6 hours
* Donor age ≥ 55 years old
* Study Center Investigator requires additional assessment ex vivo and/or extended preservation time

Donor Lung Exclusion Criteria for EVLP Assessment:

The donor lung is excluded from EVLP if at least one of the following criteria have been met:

* The donor lung has confirmed pneumonia and/or persistent purulent secretions identified via bronchoscopy
* Non-persistent purulent secretions that do not clear by hour 3 on EVLP
* The donor lung has confirmed evidence of aspiration
* The donor lung has significant mechanical lung injury or trauma
* The cold ischemic time, starting at donor aortic cross clamp/ initial flush (CIT-1), required to transport the lung from the donor site to start of the EVLP procedure at SPONSOR's facility > 10 hours

EVLP Lung Inclusion Criteria for Transplantation:

The donor lung must meet each of the following conditions post-EVLP for transplant suitability consideration by the Study Center Investigator:

* PvO2/FiO2 ≥ 350 mmHg at final EVLP evaluation time period
* and < 15% increase from baseline value (defined as the first hour collection point) to final value of pulmonary vascular resistance (PVR)
* and < 15% increase from baseline value to final value of peak airway pressure (PawP)
* and < 15% decrease from baseline value to final value of static lung compliance (Cstat)
* and the total preservation time (TPT) does not exceed the following:

  * the initial CIT-1 time from donor to EVLP > 1 hour and ≤ 10 hours
  * the EVLP time > 3 hours and ≤ 6 hours
  * the second CIT-2 from EVLP cool down to beginning of recipient implantation must be > 1 hour and ≤ 6 hours for the first lung
  * the second CIT-2 from EVLP cool down to beginning of recipient implantation must be > 1 hour and ≤ 10 hours for the second lung
* and Study Center Investigator deems lung function suitable for intended subject

EVLP Lung Exclusion Criteria for Transplantation:

The donor lung is excluded from transplant inclusion if at least one of the following criteria have been met:

* PvO2/FiO2 < 350 mmHg at final EVLP evaluation time period
* or ≥ 15% increase from baseline value to final value of pulmonary vascular resistance (PVR)
* or ≥ 15% increase from baseline value to final value of peak airway pressure (PawP)
* or ≥ 15% decrease from baseline value to final value of static lung compliance (Cstat)
* or TPT exceeds any of the following conditions:

  * CIT-1 < 1 hour or > 10 hours
  * EVLP < 3 hours or > 6 hours
  * CIT-2 < 1 hour or > 6 hours for first lung or > 10 hours for second lung
* or Study Center investigator deems lung function unsuitable for intended subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2015-07-18 (Actual); Primary Completion 2018-11-21 (Actual); Study Completion 2019-11-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Loyola University Medical Center, Chicago, Illinois
  - University of Maryland Medical Center, Baltimore, Maryland
  - University of Michigan Health System, Ann Arbor, Michigan
  - Duke University Health System, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - UPMC, Pittsburgh, Pennsylvania
  - Inova Fairfax Medical Campus, Falls Church, Virginia

REFERENCES:
- [Background] Pierre AF, Sekine Y, Hutcheon MA, Waddell TK, Keshavjee SH. Marginal donor lungs: a reassessment. J Thorac Cardiovasc Surg. 2002 Mar;123(3):421-7; discussion, 427-8. doi: 10.1067/mtc.2002.120345. PMID 11882811
- [Background] Ware LB, Wang Y, Fang X, Warnock M, Sakuma T, Hall TS, Matthay M. Assessment of lungs rejected for transplantation and implications for donor selection. Lancet. 2002 Aug 24;360(9333):619-20. doi: 10.1016/s0140-6736(02)09774-x. PMID 12241936
- [Background] Orens JB, Boehler A, de Perrot M, Estenne M, Glanville AR, Keshavjee S, Kotloff R, Morton J, Studer SM, Van Raemdonck D, Waddel T, Snell GI; Pulmonary Council, International Society for Heart and Lung Transplantation. A review of lung transplant donor acceptability criteria. J Heart Lung Transplant. 2003 Nov;22(11):1183-200. doi: 10.1016/s1053-2498(03)00096-2. No abstract available. PMID 14585380
- [Background] Kawut SM, Reyentovich A, Wilt JS, Anzeck R, Lederer DJ, O'Shea MK, Sonett JR, Arcasoy SM. Outcomes of extended donor lung recipients after lung transplantation. Transplantation. 2005 Feb 15;79(3):310-6. doi: 10.1097/01.tp.0000149504.53710.ae. PMID 15699761
- [Background] Christie JD, Carby M, Bag R, Corris P, Hertz M, Weill D; ISHLT Working Group on Primary Lung Graft Dysfunction. Report of the ISHLT Working Group on Primary Lung Graft Dysfunction part II: definition. A consensus statement of the International Society for Heart and Lung Transplantation. J Heart Lung Transplant. 2005 Oct;24(10):1454-9. doi: 10.1016/j.healun.2004.11.049. Epub 2005 Jun 4. No abstract available. PMID 16210116
- [Background] Botha P, Trivedi D, Weir CJ, Searl CP, Corris PA, Dark JH, Schueler SV. Extended donor criteria in lung transplantation: impact on organ allocation. J Thorac Cardiovasc Surg. 2006 May;131(5):1154-60. doi: 10.1016/j.jtcvs.2005.12.037. PMID 16678604
- [Background] Avlonitis VS, Wigfield CH, Golledge HD, Kirby JA, Dark JH. Early hemodynamic injury during donor brain death determines the severity of primary graft dysfunction after lung transplantation. Am J Transplant. 2007 Jan;7(1):83-90. doi: 10.1111/j.1600-6143.2006.01593.x. PMID 17227559
- [Background] Suzuki Y, Cantu E, Christie JD. Primary graft dysfunction. Semin Respir Crit Care Med. 2013 Jun;34(3):305-319. doi: 10.1055/s-0033-1348474. Epub 2013 Jul 2. PMID 23821506
- [Background] Bennett M, Horton S, Thuys C, Augustin S, Rosenberg M, Brizard C. Pump-induced haemolysis: a comparison of short-term ventricular assist devices. Perfusion. 2004 Mar;19(2):107-11. doi: 10.1191/0267659104pf729oa. PMID 15162925
- [Background] Watanabe N, Sakota D, Ohuchi K, Takatani S. Deformability of red blood cells and its relation to blood trauma in rotary blood pumps. Artif Organs. 2007 May;31(5):352-8. doi: 10.1111/j.1525-1594.2007.00392.x. PMID 17470204
- [Background] Lyu DM, Zamora MR. Medical complications of lung transplantation. Proc Am Thorac Soc. 2009 Jan 15;6(1):101-7. doi: 10.1513/pats.200808-077GO. PMID 19131535
- [Background] Cypel M, Yeung JC, Hirayama S, Rubacha M, Fischer S, Anraku M, Sato M, Harwood S, Pierre A, Waddell TK, de Perrot M, Liu M, Keshavjee S. Technique for prolonged normothermic ex vivo lung perfusion. J Heart Lung Transplant. 2008 Dec;27(12):1319-25. doi: 10.1016/j.healun.2008.09.003. PMID 19059112
- [Background] Cypel M, Rubacha M, Yeung J, Hirayama S, Torbicki K, Madonik M, Fischer S, Hwang D, Pierre A, Waddell TK, de Perrot M, Liu M, Keshavjee S. Normothermic ex vivo perfusion prevents lung injury compared to extended cold preservation for transplantation. Am J Transplant. 2009 Oct;9(10):2262-9. doi: 10.1111/j.1600-6143.2009.02775.x. Epub 2009 Aug 6. PMID 19663886
- [Background] Cypel M, Liu M, Rubacha M, Yeung JC, Hirayama S, Anraku M, Sato M, Medin J, Davidson BL, de Perrot M, Waddell TK, Slutsky AS, Keshavjee S. Functional repair of human donor lungs by IL-10 gene therapy. Sci Transl Med. 2009 Oct 28;1(4):4ra9. doi: 10.1126/scitranslmed.3000266. PMID 20368171
- [Background] Cypel M, Sato M, Yildirim E, Karolak W, Chen F, Yeung J, Boasquevisque C, Leist V, Singer LG, Yasufuku K, Deperrot M, Waddell TK, Keshavjee S, Pierre A. Initial experience with lung donation after cardiocirculatory death in Canada. J Heart Lung Transplant. 2009 Aug;28(8):753-8. doi: 10.1016/j.healun.2009.05.009. Epub 2009 Jun 28. PMID 19632569
- [Background] Yeung JC, Cypel M, Waddell TK, van Raemdonck D, Keshavjee S. Update on donor assessment, resuscitation, and acceptance criteria, including novel techniques--non-heart-beating donor lung retrieval and ex vivo donor lung perfusion. Thorac Surg Clin. 2009 May;19(2):261-74. doi: 10.1016/j.thorsurg.2009.02.006. PMID 19662970
- [Background] Cypel M, Yeung JC, Liu M, Anraku M, Chen F, Karolak W, Sato M, Laratta J, Azad S, Madonik M, Chow CW, Chaparro C, Hutcheon M, Singer LG, Slutsky AS, Yasufuku K, de Perrot M, Pierre AF, Waddell TK, Keshavjee S. Normothermic ex vivo lung perfusion in clinical lung transplantation. N Engl J Med. 2011 Apr 14;364(15):1431-40. doi: 10.1056/NEJMoa1014597. PMID 21488765
- [Background] Cypel M, Yeung JC, Keshavjee S. Novel approaches to expanding the lung donor pool: donation after cardiac death and ex vivo conditioning. Clin Chest Med. 2011 Jun;32(2):233-44. doi: 10.1016/j.ccm.2011.02.003. Epub 2011 Mar 25. PMID 21511086
- [Background] Koike T, Yeung JC, Cypel M, Rubacha M, Matsuda Y, Sato M, Waddell TK, Liu M, Keshavjee S. Kinetics of lactate metabolism during acellular normothermic ex vivo lung perfusion. J Heart Lung Transplant. 2011 Dec;30(12):1312-9. doi: 10.1016/j.healun.2011.07.014. Epub 2011 Sep 17. PMID 21930395
- [Background] Cypel M, Yeung JC, Machuca T, Chen M, Singer LG, Yasufuku K, de Perrot M, Pierre A, Waddell TK, Keshavjee S. Experience with the first 50 ex vivo lung perfusions in clinical transplantation. J Thorac Cardiovasc Surg. 2012 Nov;144(5):1200-6. doi: 10.1016/j.jtcvs.2012.08.009. Epub 2012 Aug 31. PMID 22944089
- [Background] Yeung JC, Cypel M, Machuca TN, Koike T, Cook DJ, Bonato R, Chen M, Sato M, Waddell TK, Liu M, Slutsky AS, Keshavjee S. Physiologic assessment of the ex vivo donor lung for transplantation. J Heart Lung Transplant. 2012 Oct;31(10):1120-6. doi: 10.1016/j.healun.2012.08.016. PMID 22975103
- [Background] Wigfield CH, Cypel M, Yeung J, Waddell T, Alex C, Johnson C, Keshavjee S, Love RB. Successful emergent lung transplantation after remote ex vivo perfusion optimization and transportation of donor lungs. Am J Transplant. 2012 Oct;12(10):2838-44. doi: 10.1111/j.1600-6143.2012.04175.x. PMID 23009140
- [Background] Cypel M, Keshavjee S. The clinical potential of ex vivo lung perfusion. Expert Rev Respir Med. 2012 Feb;6(1):27-35. doi: 10.1586/ers.11.93. PMID 22283576
- [Background] Munshi L, Keshavjee S, Cypel M. Donor management and lung preservation for lung transplantation. Lancet Respir Med. 2013 Jun;1(4):318-28. doi: 10.1016/S2213-2600(12)70064-4. Epub 2013 Feb 20. PMID 24429157
- [Derived] Mallea JM, Hartwig MG, Keller CA, Kon Z, Iii RNP, Erasmus DB, Roberts M, Patzlaff NE, Johnson D, Sanchez PG, D'Cunha J, Brown AW, Dilling DF, McCurry K. Remote ex vivo lung perfusion at a centralized evaluation facility. J Heart Lung Transplant. 2022 Dec;41(12):1700-1711. doi: 10.1016/j.healun.2022.09.006. Epub 2022 Sep 18. PMID 36229329

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EVLP Double Lung Group | EVLP Single Lung Group | Control Group
Started | 35 | 31 | 52
Completed | 30 | 29 | 48
Not Completed | 5 | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EVLP Double Lung Group | EVLP Single Lung Group | Control Group | Total
Number analyzed (Participants) | 35 | 31 | 52 | 118
Age, Continuous [Mean (Full Range); unit: years] | 54.9 [20 to 69] | 65.2 [55 to 72] | 61.6 [46 to 75] | 62.5 [20 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 12 | 14 | 45
  Male | 16 | 19 | 38 | 73
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 4 | 0 | 2 | 6
  White | 30 | 28 | 47 | 105
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 35 | 31 | 52 | 118
Lung Allocation Score [Mean (Full Range); unit: units on a scale] — Score developed and utilized by the United States Department of Health and Human Services to assign lung transplant waitlist priority. The score uses a combination of demographic and medical factors from each patient to assess the urgency of transplant need and the relative benefit to the patient of receiving an organ transplant.
  Refer to https://optn.transplant.hrsa.gov/resources/allocation-calculators/las-calculator/ Range of scale: 0 (zero) to 100 (one hundred). Higher numbers represent higher waitlist priority (this is not an outcome measure).
  units on a scale | 39.6 [31.1 to 69.2] | 40.0 [32.5 to 64.9] | 44.7 [31.1 to 88.5] | 42.0 [31.1 to 88.5]

OUTCOME MEASURES:

1. Primary Outcome: Count of Participants With Primary Graft Dysfunction (PGD), Grade 3
Description: Primary Graft Dysfunction is a scale published by the International Society of Heart and Lung Transplantation that uses patient oxygenation and radiographic results to score patients on a 0 (zero) to 3 (three) scale, with 3 being the most significant dysfunction.
Time Frame: 72 Hours
Measure: Count of Participants; unit: Participants
Arm/Group | EVLP Double Lung Group | EVLP Single Lung Group | Control Group
Number analyzed (Participants) | 35 | 31 | 52
Participants | 8 | 8 | 2

2. Primary Outcome: Count of Participants Surviving
Description: The number of participants that survived to 30 days post-transplant.
Time Frame: 30 Days
Measure: Number; unit: survivors
Arm/Group | EVLP Double Lung Group | EVLP Single Lung Group | Control Group
Number analyzed (Participants) | 35 | 31 | 52
survivors | 35 | 31 | 52

3. Secondary Outcome: PGD Score
Description: PGD Score (0-3) at 0, 24, 48 & 72 hours post-transplant
Time Frame: 0, 24, 48 & 72 Hours
Reporting Status: Not Posted

4. Secondary Outcome: ICU Length of Stay
Time Frame: 30 Days
Reporting Status: Not Posted

5. Secondary Outcome: Total Lung Preservation Time (TPT)
Time Frame: 72 Hours
Reporting Status: Not Posted

6. Secondary Outcome: Time to First Extubation
Time Frame: Days
Reporting Status: Not Posted

7. Secondary Outcome: Hospital Length of Stay
Time Frame: Days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Description: Regular Investigator Assessment
Arm/Group | EVLP Double Lung Group | EVLP Single Lung Group | Control Group
All-Cause Mortality (participants affected / at risk) | 5/35 | 2/31 | 4/52
Serious Adverse Events (participants affected / at risk) | 31/35 | 24/31 | 41/52
Other Adverse Events (participants affected / at risk) | 35/35 | 30/31 | 51/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EVLP Double Lung Group (N=35) | EVLP Single Lung Group (N=31) | Control Group (N=52)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 8 | 6 | 10
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 5
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6 | 4 | 7
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 6 | 4 | 4
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 2
Cytomegalovirus Viremia (Infections and infestations) | 3 | 3 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 4
Cardiac Arrest (Cardiac disorders) | 3 | 2 | 1
Lung Transplant Rejection (Immune system disorders) | 4 | 1 | 7
Delerium (Nervous system disorders) | 1 | 3 | 0
Pneumonia pseudomonal (Infections and infestations) | 2 | 2 | 0
Transplant Rejection (Immune system disorders) | 2 | 1 | 5
Septic shock (Infections and infestations) | 2 | 0 | 3
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 2 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 2 | 1
Pneumatosis intestinalis (Gastrointestinal disorders) | 3 | 0 | 0
Influenza (Infections and infestations) | 0 | 2 | 1
Postoperative wound infection (Infections and infestations) | 2 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 2 | 0 | 0
Bronchial anastomosis complication (Injury, poisoning and procedural complications) | 2 | 1 | 0
Complications of transplanted lung (Injury, poisoning and procedural complications) | 3 | 0 | 2
Cerebrovascular accident (Nervous system disorders) | 2 | 0 | 0
Syncope (Nervous system disorders) | 0 | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 2 | 1
Shock hemorrhagic (Vascular disorders) | 3 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | EVLP Double Lung Group (N=35) | EVLP Single Lung Group (N=31) | Control Group (N=52)
Atrial Fibrillation (Cardiac disorders) | 2 | 4 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 2 | 3
Dysphagia (Gastrointestinal disorders) | 1 | 2 | 1
Drug hypersensitivity (Immune system disorders) | 2 | 0 | 0
Lung transplant rejection (Immune system disorders) | 6 | 10 | 12
Transplant rejection (Immune system disorders) | 8 | 7 | 15
Bronchitis (Infections and infestations) | 3 | 0 | 1
Bronchitis bacterial (Infections and infestations) | 1 | 2 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 2 | 2 | 5
Cytomegalovirus viremia (Infections and infestations) | 1 | 2 | 3
Diverticulitis (Infections and infestations) | 1 | 2 | 0
Haemophilus infection (Infections and infestations) | 2 | 0 | 0
Infectious pleural effusion (Infections and infestations) | 2 | 0 | 0
Influenza (Infections and infestations) | 0 | 2 | 2
Lower respiratory tract infection bacterial (Infections and infestations) | 10 | 8 | 8
Lung infection pseudomonal (Infections and infestations) | 8 | 2 | 8
Pneumonia (Infections and infestations) | 1 | 3 | 3
Respiratory tract infection bacterial (Infections and infestations) | 1 | 0 | 4
Rhinovirus infection (Infections and infestations) | 1 | 2 | 5
Transmission of an infectious agent via transplant (Infections and infestations) | 2 | 1 | 4
Upper respiratory tract infection (Infections and infestations) | 3 | 1 | 1
Bronchial anastomosis complication (Injury, poisoning and procedural complications) | 1 | 2 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 2 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 2 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 3
Mental status changes (Psychiatric disorders) | 2 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0 | 0
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Decubitis ulcer (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-11-03): https://cdn.clinicaltrials.gov/large-docs/28/NCT02234128/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-08): https://cdn.clinicaltrials.gov/large-docs/28/NCT02234128/SAP_001.pdf